CLINICAL TRIAL: NCT05909293
Title: Clinical Study Protocol of Maintenance Therapy With Venetoclax in Elderly Patients With Acute Myeloid Leukemia (AML) in First Complete Remission
Brief Title: Clinical Study Protocol of Maintenance Therapy With Venetoclax in Elderly Patients With AML in First Complete Remission
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Huai'an First People's Hospital (Other); Yancheng First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-541
Record Dates: First submitted 2023-05-26; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Tablets; Granulocyte Colony-Stimulating Factor; Interleukin-11; Anti-Bacterial Agents; Antiemetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venclexta (Experimental): During the consolidation phase, which occurs within 2 months after the completion of consolidation therapy, the BCL-2 inhibitor maintenance treatment will consist of 12 cycles, with each cycle lasting 28 days.
  The specific regimen for the Venclexta is as follows:
  Venclexta: 400mg/day, orally, from day 1 to day 14 of each cycle.
  Interventions: Drug: Venclexta 100 MG Oral Tablet

INTERVENTIONS:
Drug: Venclexta 100 MG Oral Tablet — When there is a deficiency of neutrophils, G-CSF treatment may be necessary. The treatment is continued until the absolute neutrophil count (ANC) reaches either >0.5×109/L and remains at that level for 3 consecutive days, or >2×109/L. The purpose of G-CSF therapy in this context is to stimulate the production of neutrophils and restore their levels to a sufficient and stable range. This helps to strengthen the immune system and reduce the risk of infections associated with low neutrophil counts.
  When experiencing Grade 3-4 thrombocytopenia, subcutaneous injection of IL-11 can be administered as a treatment.
  When symptoms of infection occur, aggressive antimicrobial therapy and other supportive treatments should be administered.
  All blood products should undergo irradiation when transfused, and all blood products must be filtered before infusion.
  If gastrointestinal adverse reactions occur, antiemetic medications can be administered to alleviate symptoms.
  Other Names: Granulocyte colony-stimulating factor (G-CSF); Interleukin-11 (IL-11); Antibiotics; Blood products; Antiemetics

SUMMARY:
This clinical study evaluates the efficacy and safety of maintenance therapy with BCL-2 inhibitors in elderly patients with acute myeloid leukemia (AML) in first complete remission.

This study involves the following content: BCL-2 inhibitors.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, single-arm clinical study that aims to observe the efficacy and safety of maintenance therapy with BCL-2 inhibitors in elderly patients with acute myeloid leukemia (AML) in first complete remission.

The FDA has approved the combination therapy of Venetoclax and Decitabine/Azacitidine for elderly (>60 years old) newly diagnosed AML patients who are not eligible for intensive chemotherapy. Venetoclax, the first highly selective BCL-2 inhibitor available globally, is a BH3 mimetic that selectively binds to the BCL-2 protein, displacing and releasing pro-apoptotic proteins that were originally bound to BCL-2, effectively inducing apoptosis in tumor cells.

In recent years, maintenance therapy for elderly AML patients has also been under continuous exploration. In 2020, Andrew et al. published clinical trial results in the New England Journal of Medicine, demonstrating the use of oral Azacitidine formulation (CC-486) as maintenance therapy for elderly AML patients who achieved their first complete remission (CR1).

Considering the high response rate achieved by BCL-2 inhibitors in treating elderly AML and the tolerable adverse effects, maintenance therapy has shown survival benefits and good safety profiles in elderly AML patients. Therefore, your plan is to further explore, refine, and optimize treatment strategies for elderly AML patients by administering BCL-2 inhibitor maintenance therapy to those who have achieved their first CR, evaluating patient overall survival (OS), relapse-free survival (RFS), and treatment safety through a comparative study with a control group. This aims to preliminarily establish the role of this maintenance regimen in the treatment of elderly AML.

Participants will be recruited within 24 months from the completion of consolidation therapy, and the BCL-2 inhibitor maintenance therapy will last for 12 cycles, with each cycle consisting of 28 days. The analysis will be conducted approximately 48 months after the enrollment of the first patient and the follow-up will continue for 2 years from the randomization of the last patient.

Specific protocol:

During the consolidation phase, which occurs within 2 months after the completion of consolidation therapy, the BCL-2 inhibitor maintenance treatment will consist of 12 cycles, with each cycle lasting 28 days.

The specific regimen for the BCL-2 inhibitor is as follows:

BCL-2 inhibitor: 400mg/day, orally, from day 1 to day 14 of each cycle.

The target is to enroll 100 eligible patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myeloid leukemia (AML) diagnosed based on bone marrow morphology and immunophenotyping (meeting the diagnostic criteria of WHO 2016).
* Achieving first complete remission (CR) or incomplete complete remission (CRi) after 1-2 cycles of induction therapy and receiving consolidation treatment for at least 4 cycles.
* Age between 60 and 85 years.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3 times the upper limit of normal (ULN), serum bilirubin ≤ 1.5 times ULN, serum creatinine ≤ 2.0 times ULN, and serum creatine kinase < 2.0 times ULN.
* Left ventricular ejection fraction (LVEF) ≥ 50% as determined by echocardiography.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-3. Obtaining informed consent from the patient or their legal representative.

Exclusion Criteria:

* Acute promyelocytic leukemia, myeloid sarcoma, blast phase of chronic myeloid leukemia.
* Patients who achieve CR after relapse and re-induction therapy.
* Extramedullary involvement of AML, including active central nervous system leukemia.
* Allergy to any of the drugs involved in the protocol. Pregnant or lactating women and reproductive-age patients who are unwilling to use contraception.
* Significant abnormalities in liver or kidney function beyond the inclusion criteria.
* Presence of organic heart disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction with clinical symptoms or cardiac dysfunction within the past 6 months (according to New York Heart Association functional classification NYHA ≥ 3).
* Concurrent presence of other malignant tumors, except for the following conditions:

  1. Patients who have received curative-intent treatment and have not had any known active disease of malignant tumors for ≥ 5 years before enrollment.
  2. Patients who have received adequate treatment and do not show signs of disease for non-melanoma skin cancer or malignant melanocytic nevi (even if it is within 3 years before randomization).
  3. Patients who have received adequate treatment and do not show signs of disease for in situ carcinoma (even if it is within 3 years before randomization).
* Patients with HIV/AIDS, syphilis, active hepatitis B (detectable HBV-DNA), and hepatitis C.
* Any concurrent medical condition or disease (such as active systemic infection) that may interfere with the study procedures or results or pose risks to the participant as determined by the investigator.Inability to understand or comply with the study protocol.
* Patients younger than 60 years or older than 85 years.
* Undergoing major surgery within 4 weeks prior to randomization.
* Patients who have undergone allogeneic hematopoietic stem cell transplantation.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival (OS) | From the time of CR/CRi to time for up to 2 years
  2-year overall survival (OS) refers to the percentage of patients who are alive 2 years after a certain event or treatment.The time from diagnosis to patient death or the end of follow-up is calculated.
Recurrence-free survival (RFS) | From the time of CR/CRi to time for up to 2 years
  The term "Recurrence-free survival (RFS)" refers to the period of time starting from the point of complete remission (CR) or incomplete complete remission (CRi) and ending at the occurrence of leukemia relapse or any event leading to death. During this period, the patient does not experience a relapse or progression of leukemia and does not die from other causes. RFS is an important measure of survival used to assess the effectiveness of treatment in controlling leukemia relapse.

SECONDARY OUTCOMES:
Assessment of efficacy. | At the end of the 6 cycle of treatment, which corresponds to 28 days per cycle.
  CR definition: Bone marrow blast percentage less than 5%, no Auer rods, no evidence of extramedullary leukemia, peripheral blood neutrophil count greater than 1×10^9/L, and platelet count greater than 100×10^9/L. The time for hematologic recovery after induction therapy is calculated from the first day of chemotherapy.
  CRi definition: Meets all CR criteria except for ANC < 1×10^9/L or platelet count < 100×10^9/L.
  Relapse definition: Reappearance of leukemia cells in the peripheral blood after achieving CR, or bone marrow blast percentage > 5% (excluding other causes such as bone marrow regeneration after consolidation therapy), or extramedullary leukemia cell infiltration.
The impact of maintenance therapy on minimal residual disease (MRD) kinetics. | From the time of CR/CRi to time for up to 2 years
  Definition of minimal residual disease (MRD): The presence of residual leukemia cells below the threshold detected by conventional morphological methods. In this study, MRD was assessed using second-generation sequencing (NGS), real-time quantitative PCR, and multiparameter flow cytometry techniques.
Safety evaluation | From the time of CR/CRi to time for up to 2 years
  Adverse reactions will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, which provides grading standards for acute and subacute toxicities of anticancer drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China